CLINICAL TRIAL: NCT03365986
Title: Systemic Screening of Germline Cancer Gene Mutation for Colorectal Cancer in China: A Prospective and Multi-center Study
Brief Title: Systemic Screening for Hereditary Colorectal Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, professor, Sun Yat-sen University
Other Study IDs: 2017-FXY-075
Record Dates: First submitted 2017-11-26; First posted 2017-12-08 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Hereditary Colorectal Cancer
Keywords: hereditary; colorectal cancer; screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood retained, DNA was extracted for sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: genetic screening — Patients receive genetic test to see whether they have germline cancer susceptibility gene mutations

SUMMARY:
The purpose of the this study is to determine the prevalence of germline cancer susceptibility gene mutation among Chinese population, and to find best ways to screen patients with colorectal cancer in China. To accomplish this objective, the investigators will establish a large sample database of hereditary colorectal cancer related information using multigene panel testing based on Next-Generation Sequencing.

DETAILED DESCRIPTION:
Hereditary factors play a very important role in colorectal cancer risk. Identification of the germline cancer gene mutation at the time of colorectal cancer presentation has significant implications for the patients and families, as it directs follow up and clinical options. Professional guidelines recommend patients with colorectal cancer receive a phenotype-driven genetic testing strategies. For example，Lynch syndrome was identified in 2%-4% of patients with CRC using micro-satellite instability (MSI) or DNA mismatch repair (MMR) protein immunohistochemistry (IHC) tumor testing in preselected patients for germline MMR gene testing. However, there is few of clinical characteristics or germline gene mutation data from Chinese population. With the advent of next-generation sequencing (NGS), genetic testing for hereditary CRC has shifted from phenotype-specific single gene assessment to broad panels providing simultaneous assessment of multiple genes implicated in various hereditary cancer syndromes. This study plans to screen and establish a database of 500 consecutive newly diagnosed patients with CRC using multigene panel testing based on Next-Generation Sequencing. The purpose of this study is to:

1. Determine the prevalence of hereditary colorectal cancer and spectrum of germline cancer gene mutation among Chinese population.
2. Evaluate the cost-effectiveness and optimize the design of multigene panel testing.
3. Establish a statewide screening model for hereditary colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with colorectal adenocarcinoma (all stages) patients. For individuals who are old than 70 years old should meet the revised Bethesda Guidelines or polyposis syndromes testing criteria.
2. Agree to provide related information.

Exclusion Criteria:

1. Individuals who are under the age of 18.
2. Individuals who refuse to test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with colorectal adenocarcinoma (all stages). For individuals who are old than 70 years old should meet the revised Bethesda Guidelines or polyposis syndromes testing criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hereditary colorectal cancer | 3 months
  Through genetic testing for germline cancer susceptibility gene mutations among 500 consecutive patients with colorectal cancer using multigene panel testing based on Next-Generation Sequencing

SECONDARY OUTCOMES:
cost-effect for hereditary colorectal cancer screening | 3 months
  The direct cost of multigene panel testing or the traditional phenotype-specific single gene testing for hereditary colorectal cancer were estimated, and cost-effect analysis were be done between this two strategies

CONTACTS AND LOCATIONS:
Overall Officials: Ding Peirong, MD, Study Director — Sun Yat-sen University
Locations (1):
- 651 Dongfeng Road East, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Jiang W, Li L, Ke CF, Wang W, Xiao BY, Kong LH, Tang JH, Li Y, Wu XD, Hu Y, Guo WH, Wang SZ, Wan DS, Xu RH, Pan ZZ, Ding PR. Universal germline testing among patients with colorectal cancer: clinical actionability and optimised panel. J Med Genet. 2022 Apr;59(4):370-376. doi: 10.1136/jmedgenet-2020-107230. Epub 2021 Feb 9. PMID 33563768